CLINICAL TRIAL: NCT04176289
Title: PPI-guided Postoperative Pain Therapy in the OR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2112/2019
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain
Keywords: Pupillary Pain Index; Postoperative Pain; Infrared Pupillometry; Postoperative Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded study design (participants, evaluator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI-guided pain therapy (Active Comparator): At the end of anesthesia a PPI targeted opioid pain therapy will be performed by gradual administration of piritramid in 3 mg steps up to a PPI score ≤ 3.
  Interventions: Diagnostic Test: PPI measurement
- Non-PPI-guided pain therapy (No Intervention): The amount of administered piritramid in the OR will be left to the discretion of the anesthesiologist attending the participant.

INTERVENTIONS:
Diagnostic Test: PPI measurement — The pupillary dilatation reflex (PDR), induced by a standardized noxious stimulus will be measured as Pupillary Pain Index(PPI,11-point numeric scale, 0= no pain, 10= worst pain) determined with a portable pupillometer. Patients experiencing mild or more severe pain (PPI> 3) will receive intravenous opioid titration (piritramid, 3 mg bolus steps) and PPI measurement performed before and after intravenous opioid titration.
  Arms: PPI-guided pain therapy

SUMMARY:
The study will be designed to investigate the effect of pupillary pain index (PPI)-guided compared to non-PPI-guided postoperative pain therapy, conducted immediately at the end of surgery, on total postoperative opioid consumption during the first 2 postoperative hours after elective ENT surgery.

DETAILED DESCRIPTION:
Abstract

The study will be designed to investigate the effect of pupillary pain index (PPI)-guided compared to non-PPI-guided postoperative pain therapy, conducted immediately at the end of surgery, on total postoperative opioid consumption during the first 2 postoperative hours after elective ENT surgery. Pupillometric pain measurements helps clinicians determine and administer the optimized amount of opioids and so avoids opioid-induced side effects.

Background

The evaluation of pain intensity during the immediate postoperative period in the operating room (OR) is a key factor for post interventional pain treatment. However, this evaluation may be difficult when patients are still intubated, restricted in consciousness or are showing verbal impairment due to ENT surgery. Verbally impaired patients are at increased risk of under treatment for pain.

With rising opioid consumption, the risk of postoperative side effects like nausea and vomiting, sedation with a longer recovery time or respiratory depression increases. Especially in the cohort of ENT surgery patients, where a difficult airway is regularly presented, such side effects should be avoided. A means of predicting immediate postoperative pain after surgery and the response to opiate analgesics would therefore be highly desirable.

The pupillary dilatation reflex (PDR), measured by pupillometry, has been successfully used to assess intraoperative analgesic component of anesthetic regimes and correlates with pain intensity measured on a numeric rating scale (NRS).

Aims

Primary aim of this study is to investigate if a PPI-guided opioid administration immediately postoperative in the OR leads to less opioid requirement during the first 2 postoperative hours compared to a non-PPI guided treatment.

Secondary aim is to evaluate postoperative pain during the first 2 postoperative hours in patients after PPI-guided versus non-PPI guided opioid therapy in the OR.

Hypotheses

The investigators hypothesis that through a targeted pain therapy based on the measurement of immediate postoperative PPI score, opioid consumption and pain intensity can be reduced during the first 2 postoperative hours.

Methods

The study will be done by observing postoperative pain intensity using pupillometry in patients scheduled for elective ENT surgery, carrying out pain intervention (opioid therapy) and re-observing to verify the effectiveness of the targeted postoperative opioid administration in the OR. Pain on an 11-point verbal Likert response score and total opioid consumption will be recorded by a blinded investigator at 30-minute intervals for the initial 2 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-II
* able to read and understand the information sheet and to sign the consent form
* being scheduled for elective ENT surgery under general anesthesia
* age≥18 years

Exclusion Criteria:

* ASA physical status of III and above
* previous history of either drug or alcohol abuse
* difficulty to understand pain scoring system
* chronic users of analgesics or had used opioids within 12 h before surgery
* implanted electronic medical devices
* ophthalmologic diseases
* rapid sequence induction (RSI)
* psychiatric or mental disorders
* surgical procedure warranting elective postoperative ventilation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | first 2 postoperative hours
  cumulative opioid consumption within first 2 postoperative hours

SECONDARY OUTCOMES:
Postoperative Pain | first 2 postoperative hours
  Pain on an 11-point verbal Likert response score (VAS score) recorded by a blinded investigator at 30-minute intervals for the initial 2 postoperative hours. The 11-point numeric scale ranges between 0, meaning no pain, and 10, meaning worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria